CLINICAL TRIAL: NCT05936827
Title: Gyrocardiography- A New Non-invasive Cardiac Measurement Method to Measure Exercise Capacity and Cardiorespiratory Fitness
Status: Completed | Type: Observational
Sponsor: Precordior Ltd (Industry)
Collaborators: Paavo Nurmi Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: Sport Study
Record Dates: First submitted 2023-06-16; First posted 2023-07-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- athletic group: Moderate to high PA levels according to IPAQ.
  Interventions: Diagnostic Test: Ergospirometry
- non-athletic group: Low levels of PA according to IPAQ.
  Interventions: Diagnostic Test: Ergometry

INTERVENTIONS:
Diagnostic Test: Ergometry — Maximal exercise test is performed on a cycle ergometer (Ergoline 800 s; VIASYS Healthcare, Germany). The test begins at a workload of 50 W, which is increased by 25 W (males) every 1 min or the test begins with 25 W which is increased by 25 W (females) every 1 min until exhaustion.
  The mean workload during the last 4 min of work is calculated and the VO2max is estimated according to the American College of Sports Medicine (American College of Sports Medicine.
  ACSM's guidelines for exercise testing and prescription. Sixth edition. Baltimore: Williams & Wilkins 2000:304). Blood lactate concentration is measured immediately and 1 min after exhaustion from capillary samples (Biosen C-Line Glucose and Lactate analyzer, EKFdiagnostic GmbH, Germany). (Pahkala et al. 2013.)
  Groups: non-athletic group
Diagnostic Test: Ergospirometry — VO2max is measured using a stationary bicycle ergometer (Ergoline 800 s; VIASYS Healthcare, Germany. For males, the test starts with 100 W which is increased by 25 W every 1 min until volitional exhaustion. For females, the test starts with 50 W which is increased by 25 W every 1 min until volitional exhaustion.
  Ventilation and gas exchange (Vyntus CPX, Vyaire Medical Gmbh, Leibnizstrasse, Hoechberg, Germany) are measured during the test. Subject's blood lactate concentration is measured from capillary samples immediately and 1 min after exhaustion (Biosen C-Line Glucose and Lactate analyzer, EKF-diagnostic GmbH, Germany). The heart rate of the participants is followed continuously (CardioSoft GE, CardioSoft V6.51; GE Medical Systems Information Technologies, USA). (Heiskanen et al. 2021.)
  Groups: athletic group

SUMMARY:
The goal of this study is to produce a solution to measure the cardiorespiratory fitness (CRF), which can be used by commercially available smartphones without extra equipment, add-ons and special know-how.

This observational study with follow-up is to test the feasibility of a new non-invasive cardiac measurement method (gyrocardiography, GCG) in detecting hemodynamic parameters to measure exercise capacity and cardiorespiratory fitness in healthy subjects.

The objective is to produce a solution which can be used to measure the exercise capacity and cardiorespiratory fitness (CRF) of the exercisers, keep-fit athletes and professional athletes using hemodynamic parameters such as:

* Heart rate and Heart rate variability
* Cardiac Strength profile
* Systolic and diastolic phase
* Breathing frequency
* VO2max

Participants are either athletes or non-athletic persons. The athletes will perform spiroergometry and non-athletic persons ergometry to measure the CRF expressed as VO2max.

Following parameters will be measured during the (spiro)ergometry:

* Maximum workload (W)
* VO2max (ml/kg/min)
* HRmax
* Blood lactate
* Respiratory exchange ratio RER (VO2/VCO2)

The GCG measurements for acquiring the hemodynamic parameters are performed before and after the (spiro)ergometry using smartphone. During a 1- minute GCG measurement, the smart phone is placed on the chest in the middle of the sternum.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* No diagnosed cardiovascular diseases (mild hypertension or hypercholesterolemia are still allowed)
* No medication affecting heart rate (i.e. Beta blocker)
* Signed informed consent

Follow-up visit:

* Belong to non-athletic group
* Intention to change physical activity habits
* Willing to participate to the follow-up visit

Exclusion Criteria:

* Not meeting inclusion criteria
* Declined to participate
* Resting RR before the ergometry > 180/110mmHg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects from the area of Turku. Half of the subjects (n=100) are allocated to athletic group (moderate to high Physical activity, PA, levels according to International Physical Activity Questionnaire, IPAQ) and other half (n=100) to non-athletic group (low levels of PA according to IPAQ).
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The maximum (max) rate (V) of oxygen (O₂) your body is able to use during exercise. | 4 minutes
Gyrocardiography measurement | 1 minute
  Lasts 1 minute and is performed at least once at rest before the (spiro)ergometry.
Gyrocardiography measurement | 3 minutes
  Lasts 1 minute and is performed 3 minutes after the (spiro)ergometry.

SECONDARY OUTCOMES:
Heart rate per minute and Heart rate variability | 1 minute
  Lasts 1 minute and is performed at least once at rest before the (spiro)ergometry.
Heart rate per minute and Heart rate variability | 3 minutes
  Lasts 1 minute and is performed 3 minutes after the (spiro)ergometry.
Systolic and diastolic phase (blood pressure RR) | 1 minute
  Will be performed at least once at rest before the (spiro)ergometry.
Respiration rate per minute | 1 minute
  Lasts 1 minute and is performed at least once at rest before the (spiro)ergometry.
Respiration rate per minute | 3 minutes
  Lasts 1 minute and is performed 3 minutes after the (spiro)ergometry.
Cardiac Strength profile | 1 minute
  Lasts 1 minute and is performed at least once at rest before the (spiro)ergometry.
Cardiac Strength profile | 3 minutes
  Lasts 1 minute and is performed 3 minutes after the (spiro)ergometry.

CONTACTS AND LOCATIONS:
Overall Officials: Olli Heinonen, PhD, Principal Investigator — Paavo Nurmi Center
Locations (1):
- Paavo Nurmi Center, Turku, Finland